CLINICAL TRIAL: NCT02274259
Title: Randomized Trial Comparing Injection Frequency Between Aflibercept and Ranibizumab in Patients With Central Retinal Vein Occlusion With a Treat and Extend Algorithm
Brief Title: Comparing Injection Frequency Between Aflibercept and Ranibizumab in Patients With CRVO With a Treat& Extend Regimen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anders Kvanta (Other)
Responsible Party: Sponsor-Investigator, Anders Kvanta, Principal investigator, St. Erik Eye Hospital
Organization: St. Erik Eye Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 690110
Record Dates: First submitted 2014-10-02; First posted 2014-10-24 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Central Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — aflibercept; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aflibercept (Active Comparator): Aflibercept injection is given at every visit. Time to next treatment according to presence of macular edema
  Interventions: Drug: Aflibercept
- Ranibizumab (Active Comparator): Ranibizumab injection is given at every visit. Time to next treatment according to presence of macular edema
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Aflibercept — Aflibercept injection is given at every visit. Time to next treatment according to presence of macular edema
  Other Names: Eylea
  Arms: Aflibercept
Drug: Ranibizumab — Ranibizumab injection is given at every visit. Time to next treatment according to presence of macular edema
  Other Names: Lucentis
  Arms: Ranibizumab

SUMMARY:
Comparing ranibizumab and aflibercept in a treat and extend algorithm evaluating the number of needed injections over a 18 month period in patients with newly diagnosed CRVO.

DETAILED DESCRIPTION:
Forty patients diagnosed with a new central retinal vein occlusion (CRVO) of a maximum duration of 6 months will be recruited to the study. Patients will be randomized 1:1 to treatment with aflibercept ot ranibizumab.

all patients will receive 3 initial monthly injections. There after injections will be given att every visit according to a treat and extend schedule. If no macular edema is seen on the Ocular coherent tomography (OCT) examination the next treatment will be after 6 weeks. If the macula is dry after 6 weeks a new injection is given and the next visit is scheduled for another 8 weeks. If edema is seen on the OCT after 8 weeks the time to next injection is reduced to 6 weeks. Patients cannot receive an injection more often than every 4 weeks. All patients will receive an injection at least every 12 weeks.

Primary outcome: the number of needed injections over a 18 month period comparing ranibizumab and aflibercept.

Secondary outcome: Change in visual acuity, change in macular thickness. A subgroup of patients will also be evaluated with OCT angiography. A possible relationship between the Visual acuity and the foveal avascular zone will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* CRVO - naive patients, disease duration maximum 12 months, Best corrected visual acuity : 23-73 letters (20/40 - 20/320), Macular edema > 300 μm (Cirrus)

Exclusion Criteria:

* Neovascular Glaucoma Any previous treatment for CRVO. Intraocular surgery during the previous 3 months. Vascular retinopathy of other causes. Glaucoma with uncontrolled IOP (intra ocular pressure) Myocardial infarction or stroke during the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The number of needed injections over a 18 month period comparing ranibizumab and aflibercept. | 18 months

SECONDARY OUTCOMES:
Change in visual acuity | 18 months
  Change in visual acuity in ETDRS (Early Treatment Diabetic Retinopathy Study) letters
Change in macular thickness | 18 months
  Change in macular thickness measured by Cirrus OCT (µm)

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Westman, Study Chair — Study coordinator
Locations (1):
- St Eriks Eye Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Casselholmde Salles M, Kvanta A, Amren U, Epstein D. Optical Coherence Tomography Angiography in Central Retinal Vein Occlusion: Correlation Between the Foveal Avascular Zone and Visual Acuity. Invest Ophthalmol Vis Sci. 2016 Jul 1;57(9):OCT242-6. doi: 10.1167/iovs.15-18819. PMID 27409478